CLINICAL TRIAL: NCT01477931
Title: An Open-Label, 8-week Trial of Bupropion Hydrochloride Extended Release (Wellbutrin XL®) In Patients With Major Depressive Disorder (MDD) With Atypical Features.
Brief Title: Interventional Study of Wellbutrin XL in Major Depressive Disorder With Atypical Features
Acronym: WellbutrinXL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chi-Un Pae (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Chi-Un Pae, Chi-Un Pae MD, phD, Department of Psychiatry, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114003
Record Dates: First submitted 2011-11-16; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Depressive Disorder, Major
Keywords: Bupropion hydrochloride extended release; Wellbutrin XL; Major Depressive Disorder with Atypical Features
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wellbutrin XL (Experimental)
  Interventions: Drug: Bupropion extended release

INTERVENTIONS:
Drug: Bupropion extended release — 300mg once a daily, PO, 8weeks
  Other Names: Wellbutrin XL

SUMMARY:
The aims of this study are 1) to examine the clinical utility of bupropion hydrochloride extended release (Wellbutrin XL®) in patients with Major Depressive Disorder (MDD) with atypical features; 2) to evaluate the tolerability of bupropion hydrochloride extended release (Wellbutrin XL®) in patients with MDD with atypical features.

DETAILED DESCRIPTION:
Whether bupropion hydrochloride extended release (Wellbutrin XL®) improved atypical depressive symptoms has not been investigated. The investigators assumed that bupropion hydrochloride extended release (Wellbutrin XL®) will be effective and tolerable in the treatment of atypical depression in MDD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 20 years
* DSM-IV episode of MDD non-psychotic with atypical features characterized by mood reactivity and 2 or more symptoms of vegetative reversal (including overeating, oversleeping, severe fatigue or leaden paralysis, and a history of rejection sensitivity)
* More than 19 score on the 29-item HAM-D
* Ability to give informed consent

Exclusion Criteria:

* Bipolar depression
* Any Axis I psychotic disorder
* A history of suicide attempt, self-injurious action (excluding action with no intention of suicide) or overdosage (excluding apparently accidental overdosage)
* Patients with more than 3-point score of suicide (HAM-D-29 Item 18) or patients whose C-SSRS assessment suggests that they are or have been at significant risk for harming themselves or have actually harmed themselves, or who, in the opinion of the investigator (sub-investigator), are at significant risk for harming self or others
* A history of substance abuse in the previous 12 months
* A history of hypersensitivity to bupropion or any other components of the preparations used in the study (Wellbutrin SR 150mg and Wellbutrin XL 300 mg tablets)
* Serious or unstable medical disorders
* Starting or terminating psychotherapy during the previous 12 weeks,
* ECT treatment in the previous 3 months
* Subject has a life time diagnosis of anorexia nervosa or bulimia within the past 12 month
* Subject has a current or history of seizure disorder or brain injury (traumatic or disease-related) or any condition which predisposes to seizure- subject treated with other medications or treatment regimens that lower seizure threshold- subject undergoing abrupt discontinuation of alcohol or sedatives
* Subjects that previously failed adequate courses of pharmacotherapy from two different classes of antidepressants or previous adequate course(s) of bupropion
* Pregnancy or planning pregnancy - when a patient is in active reproductive age, he or she has to agree to use relevant contraception during the study
* Patients on monoamine oxidase inhibitors (MAOIs)
* Patients being treated with any other preparations containing bupropion as the incidence of seizures is dose dependent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
HAM-D-29 scores(Hamilton Depression Rating Scale 29) | 8 weeks
  Changes in HAM-D-29 scores from baseline to the end of treatment.

SECONDARY OUTCOMES:
8-atypical items on the HAM-D-29 | 8 weeks
  8-atypical items on the HAM-D-29 from baseline to end of treatment.
Tolerability | 8 weeks
  Tolerability evaluations will be determined by TEAEs(treatment-emergent adverse events) and vital signs recording.
CGI-I score(Clinical Global Impression Improvement score) | 8 weeks
  CGI-I score of 1 or 2 (proportion of the patients achieving this point at the end of treatment) or changes in total scores on CGI-S
SDS(Zung Self-Rating Depression Scale) | 8 weeks
  Change of SDS from baseline to end of treatment.
C-SSRS(The Columbia-Suicide Severity Rating Scale, changes in behaviours and ideation) | 8 weeks
  Change of C-SSRS from baseline to end of treatment.
ESQ(Epworth Sleepiness Questionnaire) | 8 weeks
  Change of ESQ from baseline to end of treatment.
Response | 8 weeks
  Response will be defined as 50% or greater reduction in HAM-D-29 scores from baseline to end of treatment.
Remission | 8 weeks
  Remission will be defined as a HAM-D-29 score of ≤ 7.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Un Pae, MD, Principal Investigator — Department of Psychiatry, Bucheon St.Mary's Hospital
Locations (6):
- South Korea (6):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Bucheon St.Mary's Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea, St.Vincent Hospital, Suwon, Gyeonggi-do
  - The Catholic University of Korea, Uijeongbu St. Mary'S Hospital, Uijeongbu-si, Gyeonggi-do
  - dongguk university MEDICAL CENTER, Kyungju, Kyoung-Book
  - Kyung Hee University Hospital, Seoul, Seoul